CLINICAL TRIAL: NCT06023251
Title: Does the Use of Supplemental Parenteral/Enteral Nutrition and/or Oral Nutrition Supplements Guided by Indirect Calorimetry Combined With Standard of Care Increases Energy Feeding Adequacy in Patients Who Survived Critical Illness?
Brief Title: Improving Nutritional Adequacy of ICU Survivors in a Prospective Interventional Way: the Bright Side Study
Acronym: BrightSide
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Elisabeth De Waele, Head of Department, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EC-2023-236
Record Dates: First submitted 2023-08-18; First posted 2023-09-05 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort (Other): oral food, enteral nutrition, parenteral nutrition
  Interventions: Other: Clinical Nutrition

INTERVENTIONS:
Other: Clinical Nutrition — Nutritional care plan implementation, including
  * A step-up and step-down nutritional protocol guided by caloric and protein ratio
  * Monitoring plan including daily nutritional intake assessment by a dietician and (para)medical supervision by a nutrition support pharmacist and nurse concerning dysphagia, refeeding syndrome, electrolytes abnormalities and access issues
  * Indirect calorimetry measurements to assess metabolic needs and body impedance analysis to assess body composition on regular time points
  * Dedicated and specialized dietician and nurse involvement
  * Adaptive communication policy (translating to native language) and culturally appropriate food regimens and artificial nutrition.

SUMMARY:
The objective is to increase caloric adequacy in patients who survived critical illness and are admitted to the ward by the use of a pro-active inclusive nutritional strategy including supplemental parenteral and/or enteral nutrition and/or oral nutritional supplements guided by indirect calorimetry.

This enables the investigators to address, within a clinical/scientific context, a recently demonstrated but until now relatively neglected 'dark side' of patient care at UZ Brussel, comparable to limited global evidence : iatrogenic malnutrition of ICU survivors. The use of a newly developed clinical pathway and nutrition strategy (oral, enteral and parenteral) led by a single SPoC (Single Point of Contact) for patients surviving intensive care will have a clear objective: to address the nutritional deficit in all patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years
* ICU stay ≥ 7 days
* Ward stay ≥ 3 days
* Nutritional therapy not restricted
* Heterogeneous diseases

Exclusion Criteria:

* Patients < 18 years
* ICU < 7 days
* Ward stay < 3 days
* Advanced Care Planning with impact on nutritional therapy
* Patients with palliative care
* Metabolic derangements such as metabolic diseases
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Nutrition Adequacy | The adequacy will be calculated over the entire ward stay: from date of inclusion till 28 days later or death from any cause, whichever came first.
  Increase of caloric adequacy (from 58 to 80%) and protein adequacy (from 52 to 80%) in ICU survivors

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth De Waele, MD PhD, Principal Investigator — Universitair Ziekenhuis Brussel, Vrije universiteit Brussel
Locations (1):
- UZ Brussel, Brussels, Belgium